CLINICAL TRIAL: NCT03835052
Title: Quality of Life Assessment in Cancer Survivors Integrated Into Routine Clinical Care Implementation in an Integrated Health System
Brief Title: QOL Assessment in Cancer Survivors Integrated Into Routine Clinical Care
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Christian S. Adonizio, MD, Medical Director: Center for Oncology Research and Innovation, Geisinger Clinic
Other Study IDs: 2018-0568
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Cancer
Keywords: Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational cohort study of patients who received cancer treatment (of any modality) in the last 18 months are evaluated by the use of a validated QOL tool (FACT-GP) and are evaluated via telephone or in person or both. Patients with high-risk for unmet needs or distress as determined by the FACT-GP are referred to an in-person Multidisciplinary Cancer Survivorship Clinic. This is considered standard of care at the investigator's institution and is part of the continuous clinical quality improvement program within the Geisinger Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignancy in the last 18 months, treated with curative intent

Exclusion Criteria:

* Patients treated with palliative intent, metastatic disease at the time of diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients meeting criteria identified through the use of analytics querying the central data architecture of health system
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Survivorship Care Plan (SCP) is completed and given to the patient | Within 12 months of date of diagnosis
  A completed Survivorship Care Plan (SCP) as defined by the American College of Surgeons, Committee on Cancer (ACS-CoC) is completed by a member of the clinical care team and is provided personally to the patient.

SECONDARY OUTCOMES:
Oncology Behavioral Health Referral Follow-up | Within 30 days of administration of FACT-GP
  FACT-GP v.4, Emotional Well-Being Sub-score (EWB) are referred to the Oncology Behavioral Health Service for an evaluation by a PhD behavioral health practitioner.
Emergency Department utilization, 30 days after completion of SCP | Within 30 days of receipt of Supportive Care Plan
  Percentage of patients who present to an Emergency Department as captured in central clinical data architecture

OTHER OUTCOMES:
Multidisciplinary Cancer Survivorship Clinic Utilization | Within 30 days of administration of FACT-GP
  Patients who have a total score less than 60 on FACT-GP are referred to the Multidisciplinary Cancer Survivorship Clinic for in-person evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Adonizio, MD, Study Chair — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No